CLINICAL TRIAL: NCT01713283
Title: A Phase 2, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Sofosbuvir Plus Ribavirin Administered for Either 12 or 24 Weeks in Treatment-Naive and Treatment-Experienced Egyptian Adults With Chronic Genotype 4 HCV Infection
Brief Title: Sofosbuvir Plus Ribavirin in Treatment-Naive and Treatment-Experienced Egyptian Adults With Chronic Genotype 4 Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0114
Expanded Access: NCT01779518 (Approved for marketing)
Record Dates: First submitted 2012-10-17; First posted 2012-10-24 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOF+RBV 12 Weeks (Experimental): Treatment-naive and treatment-experienced participants will receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (Experimental): Treatment-naive and treatment-experienced participants will receive SOF+RBV for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study is to evaluate the safety, tolerability, and antiviral activity of sofosbuvir (SOF) with ribavirin (RBV) in Egyptian adults with chronic genotype 4 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* First generation Egyptian; must have been born in Egypt and can trace both maternal and paternal Egyptian ancestry
* Treatment-experienced or treatment-naive
* Chronic genotype 4 HCV infection
* Not co-infected with HIV
* Screening laboratory values within defined thresholds
* Use of highly effective contraception methods
* Must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion Criteria:

* History of any other clinically significant chronic liver disease
* Pregnant or nursing female or male with pregnant female partner
* History of clinically-significant illness or any other major medical disorder that may interfere with treatment, assessment, or compliance with the protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kersey, MSc, Study Director — Gilead Sciences
Locations (1):
- Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one study site in the United States. The first participant was screened on 01 October 2012. The last participant observation occurred on 12 February 2014.
Pre-assignment Details: 76 participants were screened.
Groups:
- SOF+RBV 12 Wk: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 12 weeks
- SOF+RBV 24 Wk: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | SOF+RBV 12 Wk | SOF+RBV 24 Wk
Started | 31 | 29
Completed | 20 | 26
Not Completed | 11 | 3
Not completed — Lack of Efficacy | 10 | 2
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- SOF+RBV 12 Wk TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive (TN))
- SOF+RBV 12 Wk TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment experienced (TE))
- SOF+RBV 24 Wk TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment naive)
- SOF+RBV 24 Wk TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced)
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 12 Wk TN | SOF+RBV 12 Wk TE | SOF+RBV 24 Wk TN | SOF+RBV 24 Wk TE | Total
Number analyzed (Participants) | 14 | 17 | 14 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (12.4) | 54 (11.5) | 52 (15.6) | 57 (9.9) | 54 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9 | 1 | 19
  Male | 8 | 14 | 5 | 14 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 17 | 14 | 15 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 14 | 17 | 14 | 15 | 60
Liver Cirrhosis [Number; unit: participants]
  No | 11 | 13 | 11 | 11 | 46
  Yes | 3 | 4 | 3 | 4 | 14
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 3 | 1 | 6 | 0 | 10
    CT | 9 | 11 | 7 | 12 | 39
    TT | 2 | 5 | 1 | 3 | 11
HCV RNA (log10 IU/mL) [Mean (Standard Deviation); unit: log10 IU/mL] | 5.7 (0.59) | 6.2 (0.58) | 5.9 (0.74) | 6.1 (0.45) | 6.0 (0.61)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 7 | 4 | 8 | 7 | 26
  ≥ 800,000 IU/mL | 7 | 13 | 6 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 4 HCV infection who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV 12 Wk TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive)
- SOF+RBV 12 Wk TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment experienced)
Arm/Group | SOF+RBV 12 Wk TN | SOF+RBV 12 Wk TE | SOF+RBV 24 Wk TN | SOF+RBV 24 Wk TE
Number analyzed (Participants) | 14 | 17 | 14 | 15
percentage of participants | 78.6 | 58.8 | 100.0 | 86.7

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV 12 Wk: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks
Arm/Group | SOF+RBV 12 Wk | SOF+RBV 24 Wk
Number analyzed (Participants) | 31 | 29
percentage of participants | 0 | 3.4

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk TN | SOF+RBV 12 Wk TE | SOF+RBV 24 Wk TN | SOF+RBV 24 Wk TE
Number analyzed (Participants) | 14 | 17 | 14 | 15
percentage of participants
  SVR4 | 78.6 | 58.8 | 100.0 | 93.3
  SVR24 | 78.6 | 58.8 | 100.0 | 86.7

4. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as:
  1. Viral breakthrough: HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  2. Viral rebound: > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values, or
  3. Nonresponse: HCV RNA persistently ≥ LLOQ through 8 weeks of treatment
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk TN | SOF+RBV 12 Wk TE | SOF+RBV 24 Wk TN | SOF+RBV 24 Wk TE
Number analyzed (Participants) | 14 | 17 | 14 | 15
percentage of participants | 7.1 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
Time Frame: Up to Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Wk TN | SOF+RBV 12 Wk TE | SOF+RBV 24 Wk TN | SOF+RBV 24 Wk TE
Number analyzed (Participants) | 13 | 17 | 14 | 15
percentage of participants | 15.4 | 41.2 | 0 | 13.3

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV 12 Wk | SOF+RBV 24 Wk
Serious Adverse Events (participants affected / at risk) | 0/31 | 3/29
Other Adverse Events (participants affected / at risk) | 28/31 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Wk (N=31) | SOF+RBV 24 Wk (N=29)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Wk (N=31) | SOF+RBV 24 Wk (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Palpitations (Cardiac disorders) | 2 | 6
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 6
Nausea (Gastrointestinal disorders) | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 2
Fatigue (Gastrointestinal disorders) | 14 | 15
Irritability (Gastrointestinal disorders) | 6 | 10
Pain (Gastrointestinal disorders) | 4 | 6
Pyrexia (Gastrointestinal disorders) | 1 | 5
Malaise (Gastrointestinal disorders) | 0 | 2
Bronchitis (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 18 | 19
Dizziness (Nervous system disorders) | 5 | 9
Memory impairment (Nervous system disorders) | 2 | 3
Disturbance in attention (Nervous system disorders) | 0 | 2
Hypersomnia (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 16 | 14
Depression (Psychiatric disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 4
Dysuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 9
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years